CLINICAL TRIAL: NCT06893692
Title: Effect of Otage Exercise Program on Balance, Endurance and Motor Coordination in Pre-school Children.
Brief Title: Otago Exercise Program on Balance, Endurance and Motor Coordination in Pre-school Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR/AHS/25/Tooba Kaukab
Record Dates: First submitted 2025-03-19; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Normal Population
Keywords: Otago Exercise Program, Pre-School Children; Balance; Endurance; Motor Coordination; Physical Development

STUDY DESIGN:
Intervention Model Description: The current study will be randomized control trial, data will be collected from Pre-school of Lahore. Sample size will be 30. Inclusion criteria for the study will be both genders, 3-6 years age children and Guardians' informed consent and children were able to collaborate and engage throughout that intervention. Participants with associated orthopedics conditions, underlying genetic disorders and developmental delay will be excluded from the study. One experimental group will perform Otago Exercise Program along balance Training Exercises and the other control group will perform Balance Training exercises.Outcomes to be analyzed will be balance, endurance and motor coordination. For 12 weeks, participants in the study will undergo three sessions per week, lasting 40-45 minutes each. Tools used: Four-stage balance test, 30 Second chair stand test and Time up and down stairs test, Balance beam test.
Who Masked: Investigator
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Group A will perform the Otago Exercise Program. The training protocol consisted of ten repetitions, with a 60-second rest interval between sets. The training protocol consisted of three sessions per week for 12 weeks.
  Interventions: Other: Otago exercise program
- Controlled group (Active Comparator): Group B will perform Balance Training Exercises for 12 weeks of three sessions per week. BT included exercises such as a single-leg stance with eyes open and closed, standing on heels or toes, tandem and semi-tandem foot stance, tandem walking, walking backward and forward, and weight shifting.
  Interventions: Other: Balance Training Exercises

INTERVENTIONS:
Other: Otago exercise program — Experimental group: Group A will perform the Otago Exercise Program. The training protocol consisted of ten repetitions, with a 60-second rest interval between sets. The training protocol consisted of three sessions per week for 12 weeks.
  Arms: Experimental group
Other: Balance Training Exercises — Controlled group: Group B will perform Balance Training Exercises for 12 weeks of three sessions per week. BT included exercises such as a single-leg stance with eyes open and closed, standing on heels or toes, tandem and semi-tandem foot stance, tandem walking, walking backward and forward, and weight shifting.
  Arms: Controlled group

SUMMARY:
Balance training is crucial for preschool children's motor development and physical health. Engaging in endurance training enhances their aerobic capacity and fitness, leading to better health and the ability to sustain activities without fatigue. Early endurance development fosters lifelong physical activity habits, preventing childhood obesity and related health issues. Incorporating playful elements makes exercises engaging and age-appropriate. Regular balance training improves dynamic balance, essential for running, jumping, and sports, while reducing the risk of falls and injuries. Motor coordination training, combining balance and endurance, improves complex movement skills and spatial awareness. Adapting the Otago Exercise Program for young children addresses gaps in physical activity interventions, combating inactivity and obesity. This program aims to establish a foundation for lifelong physical activity and health by improving balance, endurance, and motor coordination.

The current study will be randomized control trial; data will be collected from Pre-school of Lahore. The sample size will be 30. Non-probability convenient sampling technique will be used. Inclusion criteria for the study will be both genders, 3-6 years age children and Guardians' informed consent and children were able to collaborate and engage throughout that intervention. Participants with associated orthopedics conditions, underlying genetic disorders and developmental delay will be excluded from the study. One experimental group will perform Otago Exercise Program (Warm-up Exercises and Strengthening Exercises) along balance Training Exercises and the other control group will perform Balance Training exercises (Single-leg stance with eyes open and closed, Standing on heels and toes, Tandem and semi tandem foot stance, Tandem walking, Walking backward and forward and Weight Shifting) Outcomes to be analyzed will be balance, endurance and motor coordination. For 12 weeks, participants in the study will undergo three sessions per week, lasting 40-45 minutes each. Tools used for data collection will be Four-stage balance test, 30 Second chair stand test and Time up and down stairs test, Balance beam test. Data will be analyzed through SPSS version 23.00.

DETAILED DESCRIPTION:
Balance training is crucial for preschool children's motor development and physical health. Engaging in endurance training enhances their aerobic capacity and fitness, leading to better health and the ability to sustain activities without fatigue. Early endurance development fosters lifelong physical activity habits, preventing childhood obesity and related health issues. Incorporating playful elements makes exercises engaging and age-appropriate. Regular balance training improves dynamic balance, essential for running, jumping, and sports, while reducing the risk of falls and injuries. Motor coordination training, combining balance and endurance, improves complex movement skills and spatial awareness. Adapting the Otago Exercise Program for young children addresses gaps in physical activity interventions, combating inactivity and obesity. This program aims to establish a foundation for lifelong physical activity and health by improving balance, endurance, and motor coordination.

The current study will be randomized control trial; data will be collected from Pre-school of Lahore. The sample size will be 30. Non-probability convenient sampling technique will be used. Inclusion criteria for the study will be both genders, 3-6 years age children and Guardians' informed consent and children were able to collaborate and engage throughout that intervention. Participants with associated orthopedics conditions, underlying genetic disorders and developmental delay will be excluded from the study. One experimental group will perform Otago Exercise Program (Warm-up Exercises and Strengthening Exercises) along balance Training Exercises and the other control group will perform Balance Training exercises (Single-leg stance with eyes open and closed, Standing on heels and toes, Tandem and semi tandem foot stance, Tandem walking, Walking backward and forward and Weight Shifting) Outcomes to be analyzed will be balance, endurance and motor coordination. For 12 weeks, participants in the study will undergo three sessions per week, lasting 40-45 minutes each. Tools used for data collection will be Four-stage balance test, 30 Second chair stand test and Time up and down stairs test, Balance beam test. Data will be analyzed through SPSS version 23.00

ELIGIBILITY:
Inclusion Criteria:

* Both Genders.
* 3-6 years age
* Guardian's informed consent and, children were able to collaborate and engage throughout the intervention.
* Flamingo test score between 15-30 seconds.

Exclusion Criteria:

* Associated orthopedics conditions.
* Underlying genetic disorders
* Developmental Delay

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2025-06-08 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Balance | Baseline, 3 weeks, 6 weeks, 9 weeks and 12 weeks.
  The Beam Balance Test is an effective assessment for measuring balance and stability, especially in children and older adults. Participants stand on a slightly elevated narrow beam, typically made of wood or metal, and attempt to maintain balance for 30 seconds to 1 minute. This test helps identify balance skills and potential issues.
Endurance | Baseline, 3 weeks, 6 weeks, 9 weeks and 12 weeks.
  The purpose of this test is to assess leg strength and endurance. The equipment needed includes a chair with a straight back without arm rests and a stopwatch. During the test, the participant sits in a chair with arms crossed over the chest and feet flat on the floor.
Coordination | Baseline, 3 weeks, 6 weeks, 9 weeks and 12 weeks.
  The Time Up and Down Stairs Test measures cardiovascular endurance and mobility by timing how quickly an individual can ascend and descend a set of stairs.

CONTACTS AND LOCATIONS:
Overall Officials: Tooba Kaukab, MS-PPT, Principal Investigator — Riphah International University
Locations (1):
- Muhammad Asif Javed, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hammami R, Aliani L, Gargallo P, Rebai H, Gene-Morales J, Colado JC. The effects of three types of balance training programs on measures of balance and muscle power in prepubertal children: A randomized controlled trial. J Sci Med Sport. 2023 Oct 16:S1440-2440(23)00425-5. doi: 10.1016/j.jsams.2023.10.004. Online ahead of print. PMID 39492052